CLINICAL TRIAL: NCT01241461
Title: A Phase 1 Study of LY2584702 in Japanese Patients With Solid Tumors
Brief Title: A Study of LY2584702 in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13871; I3G-JE-JGCC (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Cancer
Keywords: Advanced Cancer; Metastatic Cancer; p70s6 inhibitor
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — LY2584702

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LY2584702 (Experimental)
  Interventions: Drug: LY2584702

INTERVENTIONS:
Drug: LY2584702 — Dose escalation starting at 50 milligram (mg). On Day 1, subjects will receive a single oral dose. After a two-day observation period, subjects will receive oral doses twice daily for a 28-day cycle.
  Patients may continue 28-day cycles of twice daily dosing until discontinuation criteria are met.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of LY2584702 in Japanese patients with advanced and/or metastatic solid tumors for which no proven effective therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of a diagnosis of advanced and/or metastatic cancer (solid tumors) that is refractory to standard therapy and/or therapies known to provide clinical benefit, or for which no standard therapy exists.
* Have the presence of disease amenable to efficacy assessment as defined by the Response Evaluation Criteria In Solid Tumors (RECIST). Japanese patients who have advanced non-measurable disease with elevation of a validated tumor marker may be eligible, if discussed and agreed upon by the investigator and Lilly.
* Have adequate organ function including:

  * Hematologic: Absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/liter (L), platelets greater than or equal to 100 x 10^9/L, and hemoglobin greater than or equal to 9 gram/deciliter (g/dL) (transfusions are not allowed prior to enrollment within 2 weeks).
  * Hepatic: Bilirubin less than or equal to 1.5 times upper limit of normal (ULN), alkaline phosphatase (ALP), alanine transaminase (ALT) and aspartate transaminase (AST) less than or equal to 2.5 times ULN, or 5 times ULN for patients with hepatic metastases. Patients with bone metastases may enter with alkaline phosphatase values less than 5 times ULN, as long as other hepatic parameters meet inclusion criteria.
  * Renal: Serum creatinine less than or equal to 1.5 times ULN.
* Have a performance status of less than or equal to 2 on the Eastern Cooperative Oncology Group scale
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, cancer-related hormonal therapy prior to study enrollment and recovered from the acute effects of therapy.
* Have an estimated life expectancy of 12 weeks or greater
* Are able to swallow capsules

Exclusion Criteria:

* Have received treatment within 4 weeks of the initial dose of study drug with a drug that has not received regulatory approval for any indication.
* Have serious preexisting medical conditions or serious concomitant systemic disorders that, in the opinion of the investigator, would preclude participation in this study.
* Prior clinical history of tuberculosis (patient doubt tuberculosis is screening required), and positive test results in hepatitis B surface antigen (HBSAg), or hepatitis C antibodies (HCAb) (screening required).
* Have symptomatic central nervous system (CNS) malignancy or metastasis. Patients with treated CNS metastases are eligible provided their disease is radiographically stable, asymptomatic, and they are not currently receiving corticosteroids and/or anticonvulsants. Screening of asymptomatic patients without history of CNS metastasis is not required.
* Have hematologic malignancies, or lymphoma.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- 50 mg LY2584702: 50 milligram (mg) LY2584702 single oral dose on Day 1. After a two-day observation period, participants received oral doses twice daily for a 28-day cycle
- 75 mg LY2584702: 75 mg LY2584702 single oral dose on Day 1. After a two-day observation period, participants received oral doses twice daily for a 28-day cycle
Period: Overall Study
Arm/Group | 50 mg LY2584702 | 75 mg LY2584702
Started | 3 | 6
Completed | 0 | 0
Not Completed | 3 | 6
Not completed — Progressive Disease | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 mg LY2584702 | 75 mg LY2584702 | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.44 (7.17) | 64.07 (4.15) | 64.86 (5.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 3 | 6 | 9
Pathological Diagnosis [Count of Participants; unit: Participants]
  Adenocarcinoma, Colon | 1 | 2 | 3
  Adenocarcinoma, Esophageal | 1 | 1 | 2
  Adenocarcinoma, Gastric | 1 | 0 | 1
  Carcinoid Tumor, not otherwise specified (NOS) | 0 | 1 | 1
  Carcinoma, Esophagus | 0 | 1 | 1
  Gastrointestinal Stromal Tumors | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status Prior to Cycle 1 [Count of Participants; unit: Participants] — Classifies participants according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  Participants
    0 - Fully active | 2 | 6 | 8
    1 - Ambulatory, restricted strenuous activity | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Effects
Description: A clinically significant effect was any event that was a dose-limiting toxicity event (DLT). DLT was defined as an adverse event related to LY2584702 during Cycle 1 (Day 1 to Day 30) that fulfills any one of the following criteria; Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 or 4 non-hematological toxicity; platelet count <50.0 x 10^9/Liter (L) with bleeding; CTCAE Grade 4 platelet count decreased; neutrophil count <0.5 x 10^9/L lasting for 5 days or longer; any febrile neutropenia; CTCAE Grade 4 anemia; participant risk due to increasing toxicity.
Time Frame: Baseline through 30 days
Population: All participants who were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg LY2584702 | 75 mg LY2584702
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

2. Secondary Outcome: Number of Participants With Tumor Response
Description: Tumor response was assessed according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1. Complete Response (CR) is disappearance of all target lesions; Partial Response (PR) is ≥30% decrease in sum of longest diameter of target lesions.
Time Frame: Baseline to study completion up to Day 183
Population: All participants who were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg LY2584702 | 75 mg LY2584702
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Time Curve (AUC) of LY2584702
Description: AUC of single dose is AUC(0-12hours), and AUC of multiple doses is AUC during one dosing interval at steady state.
Time Frame: Cycle 1 Day 1: Predose, 0.5,1,2,3,5,8,12 hours; Cycle 1 Day 2:24 and 36 hours; Cycle 1 Day 3: Predose sample (before first dose on day 3); Cycle 1 Day 10: Predose,0.5,1,2,3,5,8,12 hours;Cycle 1 Day 17: Predose;Cycle 1 Day24: Predose;Cycle 2 Day 1: Predose
Population: All participants who were enrolled in the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/mL)
Groups:
- 50 mg LY2584702 Single Dose: 50 milligram (mg) LY2584702 single oral dose on Day 1
- 75 mg LY2584702 Single Dose: 75 mg LY2584702 single oral dose on Day 1
- 50 mg LY2584702 Multiple Doses: 50 mg LY2584702 oral doses twice daily for a 28-day cycle
- 75 mg LY2584702 Multiple Doses: 75 mg LY2584702 oral doses twice daily for a 28-day cycle
Arm/Group | 50 mg LY2584702 Single Dose | 75 mg LY2584702 Single Dose | 50 mg LY2584702 Multiple Doses | 75 mg LY2584702 Multiple Doses
Number analyzed (Participants) | 3 | 6 | 3 | 6
nanograms*hour/milliliter (ng*hr/mL) | 5100 (58) | 4990 (54) | 8020 (66) | 10300 (27)

4. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2584702
Time Frame: as for outcome 3
Population: All participants who were enrolled in the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | 50 mg LY2584702 Single Dose | 75 mg LY2584702 Single Dose | 50 mg LY2584702 Multiple Doses | 75 mg LY2584702 Multiple Doses
Number analyzed (Participants) | 3 | 6 | 3 | 6
nanograms/milliliter (ng/mL) | 805 (51) | 732 (56) | 1140 (78) | 1400 (47)

ADVERSE EVENTS:
Arm/Group | 50 mg LY2584702 | 75 mg LY2584702
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 mg LY2584702 (N=3) | 75 mg LY2584702 (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (5) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (3) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days